CLINICAL TRIAL: NCT04006652
Title: A Phase I Study of ApoGraft for the Prevention of Acute Graft Versus Host Disease in Haploidentical Hematopoietic Cell Transplant Recipients
Brief Title: ApoGraft for the Prevention of Acute Graft Versus Host Disease in Haploidentical Hematopoietic Cell Transplant Recipients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lost funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cellect Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201911131
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Acute Graft Versus Host Disease; Haploidentical Hematopoietic Stem Cell Transplant

STUDY DESIGN:
Intervention Model Description: The first three recipients will be treated in a sequential manner meaning that subjects will be transplanted with ApoGraft only after the engraftment of the previous subject has occurred.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Recipient (Experimental): * Will undergo institutionally standard myeloablative or reduced intensity chemotherapy or chemoradiotherapy which will be administered at the discretion of the treating physician
  * Recipients will undergo a single fresh ApoGraft transplant as per standard clinical site guidelines
  Interventions: Drug: ApoGraft
- Donor (No Intervention): -Donors will undergo apheresis from peripheral blood after daily G-CSF administration (for up to 5 days prior to Day -1)

INTERVENTIONS:
Drug: ApoGraft — ApoGraft is a cell based product, manufactured with mobilized peripheral blood.
  Arms: Recipient

SUMMARY:
Finding a donor remains a challenge for patients in need of an urgent hematopoietic stem cell transplantation (HSCT). The ability to obtain half matched stem cells from any family member represents a significant breakthrough in the field. Haploidentical haplo-HSCT is characterized by the nearly uniform and immediate availability of a donor and the availability of the donor for post-transplant cellular immunotherapy. However, haplo-HSCT has a high risk of Graft versus Host Disease (GvHD) and poor immune reconstitution when GvHD is prevented by all existing methods of vigorous ex vivo or in vivo T-cell depletion. Different treatment approaches are currently being explored to mitigate complications such as graft rejection, severe GvHD, and prolonged immune suppression. Novel experimental utilization of T regulatory cells, alloreactive natural killer (NK) cells, and other T cell subsets hold great promise. Cellect Biotherapeutics' platform technology, ApoGraft, is based on the findings that GvHD can be prevented by Fas receptor mediated selective depletion of T cell subsets, ex vivo. The investigators hypothesize that the use of ApoGrafts for haplo-HSCT will be safe, and reduce rates of GVHD without affecting Graft-versus-Leukemia (GvL).

ELIGIBILITY:
Recipient Inclusion Criteria:

* Adult male or female subjects, 18-70 years of age.
* Availability of an HLA-haploidentical-HSCT related donor with a minimum match of 5/10 at the HLA A, B, C, DR and DQ loci.
* Hematologic malignancy in remission or controlled as below:

  * Acute myelogenous leukemia (AML) and Acute lymphoblastic leukemia (ALL) in 1st or subsequent complete remission (CR)
  * Non-Hodgkin's Lymphoma (NHL) in CR by CT or PET/CT
  * Hodgkin's disease (HD) in 1st or subsequent CR by CT or PET/CT
  * Intermediate or high risk Myelodysplastic syndrome (MDS) (IPSS-R criteria)
* ECOG performance status score 0-1 at time of the screening visit
* Cardiac left ventricular ejection fraction ≥ 40% in adults within 90 days of start of lymphodepleting chemotherapy
* Pulmonary function test with DLCO, FEV1 and FVC of ≥ 50% within 90 days of start of lymphodepleting chemotherapy.
* Oxygen saturation ≥ 90% on room air at screening visit.
* Subjects must have adequate organ function as defined below within 2 weeks of Day 0:

  * AST (SGOT)/ALT (SGPT) ≤ 2.5 × upper limit of normal (ULN).
  * Serum bilirubin <3 mg/dL.
  * Estimated creatinine clearance >50
* If female of childbearing potential, agree to use an acceptable method of birth control or be surgically sterile, and have a negative pregnancy test.
* Available HLA-haploidentical donor
* Must be able to receive GvHD prophylaxis with tacrolimus, mycophenolate mofetil, and cyclophosphamide
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable). Subjects requiring a guardian to sign informed consent will not be included.

Recipient Exclusion Criteria:

* If a matched related donor is available and able to donate
* Participation in an interventional investigational trial within 30 days of Day 0.
* Subject suffering from any active or ongoing malignancy (other than the reason for HSCT) in the last 5 years prior to baseline; excluding basal cell carcinoma, in situ malignancy, low-risk prostate cancer, cervix cancer after curative therapy.
* Uncontrolled infections (bacterial, viral or fungal including sepsis, pneumonia with hypoxemia, persistent bacteremia, or meningitis within two weeks of the screening visit).
* Current known active acute or chronic infection with HBV or HCV.
* Known human immunodeficiency virus (HIV) infection or AIDS.
* Subjects with severe or symptomatic restrictive or obstructive lung disease or respiratory failure requiring ventilator support.
* Subjects with other concurrent severe and/or uncontrolled medical condition, which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, and chronic liver or renal disease)
* History of any of the following within 12 months prior to screening: Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), unstable angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism.
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder or any chronic condition susceptible, in the opinion of the investigator, of interfering with the conduct of the study.
* Organ allograft transplant recipient.
* If female of childbearing potential, agree to use an acceptable method of birth control or be surgically sterile, and have a negative pregnancy test.
* Pregnancy or lactation
* Must not have undergone a prior allogeneic donor (related, unrelated, or cord) transplant. Prior autologous transplant is not exclusionary.
* Presence of donor-specific anti-HLA antibodies.
* Must not receive antithymocyte globulin as part of pre-transplant conditioning regimen, plan to receive a T-cell depleted product, or have planned donor leukocyte infusions post-transplant.
* Immunosuppressive doses of steroids. Subjects with steroids for adrenal insufficiency will not be excluded.

Donor Inclusion Criteria

* Adult male or female subjects, 18-65 years of age.
* Donor criteria according to standard NMDP criteria for donor selection.

  * Blood-related family member (sibling (full or half), offspring, parent, cousin, niece or nephew, aunt or uncle, or grandparent).
  * HLA-haploidentical donor/recipient match by at least low-resolution typing per institutional standards.
  * In the investigator's opinion, donor is in general good health, and medically able to tolerate leukapheresis required for harvesting HSC.
* Fit to receive G-CSF and donate peripheral blood stem cells.
* Able to sign written informed consent including consent for 2nd donation in the event of graft failure in the recipient.

Donor Exclusion Criteria

* HIV, HBV or HCV positive subjects within 30 days prior to day 0.
* Pregnant or lactating women.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Graft donation with less than 0.3% CD34+ cells

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ApoGraft as measured by adverse events related to ApoGraft product | From day 0 to 1 year post-transplantation of ApoGraft product
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for all toxicity reporting.

SECONDARY OUTCOMES:
Cumulative incidence of graft failure | 35 days post haplo-HCT
  -Failure to engraft will be defined as failure to achieve absolute neutrophil count > 500 for 3 days by Day 35
Treatment related mortality | Through 1 year post-transplantation of ApoGraft product
  -Death that results from a transplant procedure-related complication (e.g. infection, organ failure, hemorrhage, GVHD) rather than from relapse of the underlying disease or an unrelated cause.
Time of neutrophil engraftment as determined by number of days for reaching first of 3 consecutive days with ANC ≥ 500/mm3 | 35 days post haplo-HCT
Rate of neutrophil engraftment as determined by number of days for reaching first of 3 consecutive days with ANC ≥ 500/mm3 | 35 days post haplo-HCT
Time of platelet engraftment determined by number of days for reaching first measurement of 3 consecutive measurements with platelets ≥ 20,000/mm3 in the absence of platelet administration during the prior 7 days | 35 days post haplo-HCT
Rate of platelet engraftment determined by number of days for reaching first measurement of 3 consecutive measurements with platelets ≥ 20,000/mm3 in the absence of platelet administration during the prior 7 days | 35 days post haplo-HCT
Incidence of Grade 2-4 acute GVHD | Day 180
  -Acute GVHD will be assessed using MAGIC criteria
Time to development of Grade 2-4 acute GVHD | Day 180
  -Acute GVHD will be assessed using MAGIC criteria
Incidence of Grade 3-4 acute GVHD | Day 180
  -Acute GVHD will be assessed using MAGIC criteria
Time to development of Grade 3-4 acute GVHD | Day 180
  -Acute GVHD will be assessed using MAGIC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu